CLINICAL TRIAL: NCT07261150
Title: Histoplasmosis Induction and Consolidation Therapy Factorial Randomized Clinical Trial (Histo-FACT)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDIM-2025-33491
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Histoplasmosis
MeSH Terms: conditions — Histoplasmosis | interventions — posaconazole; World Health Organization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Induction Therapy - Experimental (Experimental): Single high-dose (10mgkg) of LAmB B
  Interventions: Drug: LAmB B
- Induction Therapy - Standard of Care (Active Comparator): SOC daily standard dose (3mg/kg) LAmB
  Interventions: Drug: World Health Organization (WHO)-recommended SOC
- Consolidation Therapy - Experimental (Experimental): posaconazole
  Interventions: Drug: Posaconazole
- Consolidation Therapy - Standard of Care (Active Comparator): SOC itraconazole
  Interventions: Drug: WHO-recommended SOC Itraconazole
- Total Consolidation - Experimental (Experimental): 6 months total (e.g., 0 additional months) of itraconazole or posaconazole based on assignment from Aim 2.
  Interventions: Drug: Posaconazole; Drug: WHO-recommended SOC Itraconazole
- Total Consolidation - Standard of Care (Active Comparator): 12 months total (e.g., 6 additional months) of itraconazole or posaconazole based on assignment from Aim 2
  Interventions: Drug: Posaconazole; Drug: WHO-recommended SOC Itraconazole

INTERVENTIONS:
Drug: LAmB B — intravenous liposomal amphotericin B (10mg/kg)
  Arms: Induction Therapy - Experimental
Drug: Posaconazole — Posaconazole delayed-release tabs, 300mg twice daily on day 1 then once daily
  Arms: Consolidation Therapy - Experimental; Total Consolidation - Experimental; Total Consolidation - Standard of Care
Drug: World Health Organization (WHO)-recommended SOC — daily intravenous liposomal amphotericin B 3mg/kg, for 2 weeks or at least 7 days if felt stable for discharge per the clinician
  Arms: Induction Therapy - Standard of Care
Drug: WHO-recommended SOC Itraconazole — 200mg capsules three times daily x 3 days then twice daily
  Arms: Consolidation Therapy - Standard of Care; Total Consolidation - Experimental; Total Consolidation - Standard of Care

SUMMARY:
The purpose of the study is threefold:

1. Assess the safety and efficacy of a single high-dose intravenous (LAmB 10mg/kg) compared to the SOC daily dosing (3mg/kg) of the same medication for induction therapy in moderate to severe histoplasmosis.
2. Assess the safety and efficacy of oral posaconazole 300mg delayed-release tablets three times daily for two days then once daily for consolidation therapy compared to SOC oral itraconazole 200 mg capsules three times daily for three days then twice daily in moderate to severe histoplasmosis
3. Assess the safety and efficacy of 6 months of consolidation therapy compared to the SOC 12 months of consolidation therapy in persons with HIV on appropriate antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Hospitalized with suspected histoplasmosis b
* Diagnosis of confirmed or probable histoplasmosis (via positive Histoplasma antigen test, culture, histopathology or microscopy)
* Provision of Informed Consent by participant or surrogate c

Exclusion Criteria:

* Previous diagnosis of histoplasmosis
* Pregnant persons (all persons who could potentially be pregnant will have a pregnancy test prior to enrollment, and if negative, must agree to contraception for the duration of the study)
* Breastfeeding and unable to stop for the duration of the study
* Renal impairment (serum creatinine or blood urea nitrogen (BUN) >2.0x upper limit of normal)
* Allergy or contraindication to a study medicine
* More than one dose of an amphotericin product in the prior 7 days
* Suspected central nervous system involvement of histoplasmosis
* Likely to die in the next 48 hours in the judgment of the investigator
* Unlikely to follow up for the duration of the study in the judgement of the investigator
* Significant drug-drug interaction with itraconazole or posaconazole (such as rifampin in persons with TB)
* Current diagnosis of cryptococcosis or leishmaniasis
* QTc interval consistently >450 milliseconds
* Prisoners
* Unable to take oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality at 2 weeks | Week 2
Mortality at 26 weeks | Week 26
SAE-free survival between 26 and 52 weeks from induction therapy among those who survived 26 weeks | Week 52

SECONDARY OUTCOMES:
Aim 1: Hierarchical composite end point | Week 56
  Consisting of the following in a hierarchical order:
  5: Death within 10 weeks or lost to follow up in the first 1 week 4: Serious Adverse event within 10 weeks 3: Grade 4 laboratory abnormality at week two visit or discontinuation of medication due to intolerance during the first 10 weeks 2: Grade 3 laboratory abnormality at week two visit
  1: Alive at the end of the study period without one of the above events
Aim 2: Hierarchical composite end point | Week 56
  Consisting of the following in a hierarchical order:
  5: Death within the study period 4: Serious Adverse event within 26 weeks 3: Grade 4 laboratory abnormality through week 26 or discontinuation of medication due to intolerance during the first 26 weeks 2: Grade 3 laboratory abnormality through week 26 or or lost to follow up after the first week
  1: Alive at the end of the study period without one of the above events

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Bahr, MD, Principal Investigator — University of Minnesota
Locations (2):
- University of Minnesota, Minneapolis, Minnesota, United States
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No